CLINICAL TRIAL: NCT01426230
Title: A Phase 4, Open Label, Study of Safety and Effectiveness of GRALISE™(Gabapentin) Tablets in the Treatment of Patients With Postherpetic Neuralgia in Clinical Practice
Brief Title: Phase IV Study of FDA Approved, Once-Daily GRALISE™(Gabapentin) Tablets for the Treatment of Postherpetic Neuralgia
Status: Completed | Type: Observational
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Other Study IDs: 81-0067
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Post Herpetic Neuralgia
Keywords: PHN; Post Herpetic Neuralgia; Shingles; HZ roster
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Open Label: Cohort by age-
  - Patients >70 Yrs old
- Open label: Cohort by age-
  - Patients < 70 Yrs old

SUMMARY:
Study objective is to assess the safety and effectiveness of once- daily GRALISE in clinical practice

DETAILED DESCRIPTION:
Open Label, single arm, 2wk titration, 6 wk stable dosing, 8 wk of total treatment, 1wk dose tapering

ELIGIBILITY:
Inclusion Criteria:

* Men or Women 18 years or older who are suffering from PHN

Exclusion Criteria:

* Patient is Pregnant or a nursing mother
* Patient has hypersensitivity to gabapentin
* Patient has an estimated creatinine clearance of <30 mL/min or is in hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently suffering from Post Herpetic Neuralgia
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Sathyanarayana, Study Director — Depomed Clinical Operations
Locations (37):
- United States (37):
  - Mobile, Alabama
  - Tuscaloosa, Alabama
  - Phoenix, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - Fresno, California
  - San Francisco, California
  - Fairfield, Connecticut
  - Lauderdale Lakes, Florida
  - Naples, Florida
  - North Palm Beach, Florida
  - Ormond Beach, Florida
  - Palm Beach, Florida
  - Sunrise, Florida
  - Marietta, Georgia
  - Bolingbrook, Illinois
  - Evansville, Indiana
  - Lexington, Kentucky
  - Brighton, Massachusetts
  - Worcestor, Massachusetts
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Tom River, New Jersey
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Allentown, Pennsylvania
  - Altoona, Pennsylvania
  - Wyomissing, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Cordova, Tennessee
  - Austin, Texas
  - Bedford, Texas
  - Corpus Christi, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Orem, Utah
  - Edmonds, Washington

REFERENCES:
- [Derived] Mehta N, Bucior I, Bujanover S, Shah R, Gulati A. Relationship between pain relief, reduction in pain-associated sleep interference, and overall impression of improvement in patients with postherpetic neuralgia treated with extended-release gabapentin. Health Qual Life Outcomes. 2016 Apr 1;14:54. doi: 10.1186/s12955-016-0456-0. PMID 27037091

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 201 patients were enrolled, but only 197 patients received study treatment.
Groups:
- Open Label - Cohort >70 Yrs Old: Cohort by age-
  - Patients >70 Yrs old
- Open Label - Cohort <=70 Yrs Old: Cohort by age-
  - Patients <=70 Yrs old
Period: Overall Study
Arm/Group | Open Label - Cohort >70 Yrs Old | Open Label - Cohort <=70 Yrs Old
Started | 86 (90 patients were enrolled, but only 86 received study treatment.) | 111
Completed | 55 | 84
Not Completed | 31 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label - Cohort >70 Yrs Old | Open Label - Cohort <=70 Yrs Old | Total
Number analyzed (Participants) | 86 | 111 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 0 | 65 | 65
  >=65 years | 86 | 45 | 131
Age Continuous [Mean (Standard Deviation); unit: years] | 78.2 (5.28) | 59.0 (10.42) | 67.4 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 75 | 122
  Male | 39 | 36 | 75
Region of Enrollment [Number; unit: participants]
  United States | 86 | 111 | 197

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Study in LOCF VAS
Description: Change from baseline in pain score on visual analog scale (VAS) (intensity scored from "No Pain" (0mm) to "Worst Possible Pain" (100mm)) at Week 8 of treatment; last observation carried forward (LOCF) analysis
Time Frame: 8 weeks (Baseline and Week 8)
Population: The Number of Participants Analyzed was based on the available VAS.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Open Label - Cohort >70 Yrs Old | Open Label - Cohort <=70 Yrs Old
Number analyzed (Participants) | 80 | 110
scores on a scale | -20.4 [-26.5 to -14.4] | -21.3 [-26.8 to -15.8]

ADVERSE EVENTS:
Arm/Group | Open Label - Both Cohorts
Serious Adverse Events (participants affected / at risk) | 5/197
Other Adverse Events (participants affected / at risk) | 38/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label - Both Cohorts (N=197)
Coronary artery disease (Cardiac disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label - Both Cohorts (N=197)
Dizziness (Nervous system disorders) | 27 (28)
Somnolence (Nervous system disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: The PI agrees that sponsor shall have the right to the first publication of the study results which is intended to be a joint, multi-center publication. Following the first publication, the PI may publish study data or results, provided however PI submits the proposed publication to sponsor for review at least 60 days prior to the date of the proposed publication. Sponsor may remove any information that is considered confidential and/or proprietary other than study data.